CLINICAL TRIAL: NCT04920188
Title: LCCC 2103: Development and Application of a Novel Digital Array PCR Assay for Evaluation of Minimal Residual Disease in Acute Myeloid Leukemia (AML)
Brief Title: Development and Application of a Novel Digital Array PCR for Acute Myeloid Leukemia (AML)
Status: Terminated | Type: Observational
Why Stopped: Resources related issues
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 2103
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Leukemia, Myeloid, Acute; Minimal Residual Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: The purpose of this trial is to investigate whether a digital array assay can detect trace amounts of residual leukemia and predict relapse in acute myeloid leukemia (AML) patients in remission who have undergone allogeneic stem cell transplantation (SCT) at the North Carolina Cancer Hospital (NCCH).

Participants: Adult patients (18 years of age or older) with diagnosed AML who are going to undergo stem cell transplant (SCT).

Procedures (methods): A total of 10 eligible subjects will be treated per standard of care with SCT. Peripheral blood and bone marrow aspirate (10 mL each) for digital array assay analysis will be collected along with routine lab draws and bone marrow biopsy procedures prior to SCT. Beginning 1 month after SCT peripheral blood (10 ml) will be collected to assess MRD by digital array assay analysis on a monthly basis for up to 6 months. In addition, bone marrow aspirate will be collected at approximately Month 3 and 6 following SCT for assay analysis. Patient medical records will be reviewed 6 and 12 months after completing their last MRD follow up assessment to confirm survival status, remission status, and gather information related to relapse.

DETAILED DESCRIPTION:
Minimal residual disease (MRD) refers to the presence of cancer cells that are present after therapy and not otherwise detectable by clinical findings, including standard clinical assays and radiographic imaging. Detection of MRD before it becomes clinically detectable provides an opportunity to intervene and optimize treatment, with the possibility of curing more patients. For the above reasons, detection of MRD through evaluation of blood-based biomarkers represents a promising area to improve clinical outcomes in patients with a variety of solid and liquid tumors. In liquid tumors such as acute lymphoblastic leukemia (ALL), MRD assessment is already part of routine clinical practice. MRD is strongly correlated with risk for relapse in ALL, and MRD assessment during and after induction therapy is one of the most informative prognostic markers available. For these reasons the National Comprehensive Cancer Network (NCCN) Guidelines Version 2.2020, indicate that MRD assessment is an "essential component of patient evaluation over the course of sequential therapy" for ALL, and there are >250 references to MRD in the pediatric and adult ALL NCCN Guidelines. In AML, MRD assessment is routinely used in academic medical centers. MRD is also strongly associated with risk of relapse in AML, and MRD status is a strong independent predictor of overall survival after completion of therapy. The AML NCCN Guidelines Version 3.2020, indicate the "undeniable need for monitoring," but further refinements are needed to make MRD monitoring in patients with AML more reliable. In this study we will apply a new highly multiplexed digital PCR technology, digital array PCR (daPCR), for evaluation of MRD in AML that will improve MRD assay reliability while reducing costs and time-to-results.

Currently, methods for MRD assessment in AML include flow cytometry for the detection of aberrant immunophenotypes as well as molecular PCR- and next generation sequencing (NGS)-based assays for detecting recurrent AML-associated genetic abnormalities. Both flow and molecular MRD assessment have much higher sensitivity than morphologic assessment alone, with flow cytometry having a lower limit of detection between 10-4 to 10-5 and molecular methods between 10-3 for NGS methods to 10-5 for PCR-based methods. Each of the current methods have major limitations that prevent broader adoption in AML. Standard NGS-based methods have insufficient sensitivity and high costs. Flow cytometry is a technically difficult method that is challenging to standardize, and a subset of AML cases do not have sufficient evaluable surface markers to allow detection. PCR-based methods can be very sensitive, but each assay currently targets a single recurrent genetic abnormality (e.g., PML/RARA fusion in acute promyelocytic leukemia), and many AML cases do not have genetic abnormalities that are targeted by current clinical assays. In contrast, the daPCR technology we propose to apply in this study provides a high throughput, multiplexed platform (24-96 variants) with unprecedented dynamic range (>108), high ease of use, low cost and rapid turnaround time. Because the daPCR can simultaneously probe for multiple variants, we estimate that our initial assay will have the potential to detect and quantify the abundance of at least one AML associated mutation in ~80% of AML samples. This technological advance would provide a real-world solution to enable frequent, deep monitoring of therapeutic response in patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age) diagnosed with AML who are going to undergo stem cell transplant (SCT). These subjects must provide written informed consent to participate.
* Subjects must have an identified mutation that has been validated on the multiplex daPCR assay.

Exclusion Criteria:

* Adult patients (≥18 years of age) diagnosed with AML who are scheduled to undergo SCT at the NCCH who do not provide written informed consent to participate are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years of age or older) with diagnosed AML who are going to undergo stem cell transplant (SCT).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Detection of AML Specific mutations from peripheral blood | 2 years
  Signal intensity above negative control at mutation sites

SECONDARY OUTCOMES:
Proportion of AML patients with detectable mutations | 2 years
  Fraction of screened AML patients whose disease has a mutation that detectable on the first generation mutation panel.
Association between AML specific mutation and relapse at 6 months | 2 years
  Positive signal intensity and relapse information from medical recordrelapse at any time after initial detection.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Armistead, MD, Principal Investigator — UNC
Locations (1):
- North Carolina Cancer Hospital (NCCH), Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials